

#### **Informed Consent**

# INFORMED CONSENT/AUTHORIZATION FOR PARTICIPATION IN RESEARCH

An Investigator-Initiated, Phase II, Single-Center, Randomized, Open-Label, Prospective Study to Determine the Impact of Serial Procalcitonin on Improving Antimicrobial Stewardship and on the Efficacy, Safety, and Tolerability of Imipenem-Cilastatin-Relebactam Plus/Minus Vancomycin or Linezolid Versus Standard-of-Care Anti-Pseudomonal Beta-Lactams Plus/Minus Vancomycin or Linezolid as Empiric Therapy in Febrile Neutropenic Adults with Cancer

2020-0074

| The state of the s | |
|---|---|
| <b>Subtitle:</b> Phase II Single-Center, Randomiz<br>Impact of Serial Procalcitonin | zed, Open-Label, Prospective Study to Determine the |
| Study Chair: Issam I. Raad, M. | .D. |
| Participant's Name | Medical Record Number |

This is an informed consent and authorization form for a research study. It includes a summary about the study. A more detailed description of procedures and risks is provided after the summary.

This research has been reviewed and approved by an Institutional Review Board (IRB - a committee that reviews research studies).

#### STUDY SUMMARY

The goal of this clinical research study is to learn if the antibiotic combination imipenem-cilastatin-relebactam can help to control febrile neutropenia (fever due to low white blood cell counts) in patients with cancer. Imipenem-cilastatin-relebactam will be compared to the standard-of-care treatment (cefepime, meropenem, or piperacillin/tazobactam) for febrile neutropenia. The safety and tolerability of the study drug will also be studied.

This is an investigational study. Imipenem-cilastatin-relebactam is FDA approved and commercially available to treat certain types of infections. It is not approved for the treatment of febrile neutropenia. Its use in this study is for research purposes only. All other antibiotics given on this study are FDA approved and commercially available for the treatment of infections. However, only cefepime is specifically FDA

approved to treat febrile neutropenia. The study doctor can explain how the study drugs are designed to work.

The study drugs may help to control your infection/febrile neutropenia. Future patients may benefit from what is learned. There may be no benefits for you in this study.

Your participation is completely voluntary. Before choosing to take part in this study, you should discuss with the study team any concerns you may have, including side effects, hospitalization, potential expenses, and time commitment. If you take part in this study, you may be foregoing some standard approved treatment options.

You can read a list of potential side effects below in the Possible Risks section of this consent.

You may receive the study drug(s) for up to 14 days.

Imipenem-cilastatin-relebactam will be provided to you at no cost while you are on this study. You and/or your insurance provider will be responsible for any other antibiotic or drug you receive during this study.

You may choose not to take part in this study. Instead of taking part in this study, you may choose to receive vancomycin, linezolid, cefepime, meropenem, and/or piperacillin/tazobactam without taking part in this study. The study doctor can explain with other standard treatments are available and can discuss the potential risks and benefits with you. You may choose to receive other investigational therapy, if available. You may choose not to receive treatment against the infection at all. In all cases, you will receive appropriate medical care, including treatment for pain and other symptoms of infection.

#### 1. STUDY DETAILS

#### **Screening Tests**

Signing this consent form does not mean that you will be able to take part in this study. The following screening tests will be performed within 24 hours before your first dose of study drugs to help the doctor decide if you are eligible:

- You will have a physical exam.
- Blood (about 1 tablespoon) will be drawn for routine tests and to check for bacterial infection.
- Urine will be collected for routine tests.
- If the doctor thinks it is needed, you will have a chest x-ray or CT scan to check your lung function.
- If you can become pregnant, part of the above blood or urine sample will be collected for a pregnancy test. To take part in this study, you must not be pregnant.

The study doctor will discuss the screening test results with you. If the screening tests show that you are not eligible to take part in the study, you will not be enrolled. Other treatment options will be discussed with you.

### **Study Groups**

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the flip of a coin) 1 of 2 study groups. This is done because no one know if one study group is better, the same, or worse than the other group.

- If you are assigned to Group 1, you will receive imipenem-cilastatinrelebactam.
- If you are assigned to Group 2, you will receive a standard-of-care antibiotic (either cefepime, meropenem, or piperacillin/tazobactam) based on what the doctor in the emergency room (ER) thinks is best for you.

Both you and the study doctor will know which drug you are assigned to receive.

Up to 100 participants will take part in this study. All will be enrolled at MD Anderson.

#### **Study Drug Administration**

**If you are in Group 1,** you will receive imipenem-cilastatin-relebactam by vein over 30 minutes every 6 hours for at least 2 days.

If you are in Group 2, you will receive cefepime, meropenem, or piperacillin/tazobactam by vein for at least 2 days. If you receive cefepime or meropenem, you will receive it over 30 minutes every 8 hours. If you receive piperacillin/tazobactam, you will receive it over about 1 hour every 8 hours.

In both groups, after 2 days, if the study doctor thinks it is in your best interest and you are eligible, you may switch to receive a different antibiotic either by mouth or by vein. The study doctor will tell you more about what antibiotic you may receive, how it is administered, and its possible risks. If you begin taking the antibiotic by mouth, the study doctor will tell you how and when to take each drug.

You may receive antibiotics for up to 14 days, regardless of whether you stay on your assigned antibiotic or receive a different antibiotic during this study.

If the study doctor thinks it is needed, you will be given additional standard drugs (including vancomycin, daptomycin, linezolid, and/or other antibacterial therapy) to help control the infection. You may ask the study staff for information about how the drugs are given and their risks.

You will no longer be able to receive the study drugs if the disease gets worse, if intolerable side effects occur, if you need treatment that is not allowed on this study, or if you are unable to follow study directions.

#### **Study Visits**

You will have the following tests/procedures while you are in the hospital. If you begin to take the study drugs by mouth, you will no longer have these study visits.

**Each day for up to 2 weeks,** if the doctor thinks it is needed, blood (about 1 tablespoon) or urine will be collected for routine tests. On Day 7, these tests will only be done if you have a fever.

**Every 2 days for up to 2 weeks**, blood (about 1 tablespoon) will be drawn to check for infection. You will stop having these blood draws when there is no longer a sign of infection and you do not have a fever.

**Every 3 days after your first dose,** you will have a physical exam. If the study doctor thinks it is needed, this exam may be repeated.

### Follow-Up

Within 72 hours (3 days) after your last dose of assigned study treatment and before starting the second antibiotic therapy, if applicable:

- You will have a physical exam.
- Blood (about 1 tablespoon) will be drawn for routine tests.
- Urine will be collected for routine tests.
- If you tested positive for infection at the beginning of the study, blood (about 1 tablespoon) will be drawn to check for infection.

**About 21-28 days (3-4 weeks) after your first dose of study drug,** you will return to MD Anderson for the following tests/procedures:

- You will have a physical exam.
- Blood (about 1-2 teaspoons) will be drawn for routine tests.
- If you tested positive for infection at the beginning of the study, blood (about 1 tablespoon) will be drawn to check for infection.
- If the doctor thinks it is needed, urine may be collected for routine tests.
- If you can become pregnant, blood (about 1 teaspoon) will be drawn for a pregnancy test.

About 35-42 days (5-6 weeks) after your first dose of study drug, the study staff will call you to ask about any new drugs you may have started and if you are having any side effects. The phone call should take about 10 minutes. If the study doctor thinks it is needed, you may be asked to come back to the clinic for the following tests/procedures:

- You will have a physical exam.
- If the doctor thinks it is needed, blood (about 1 tablespoon) will be drawn to check for infection.
- If the doctor thinks it is needed, urine may be collected for routine tests.

At any of these follow-up visits, if your doctor thinks it is needed, you may have a chest x-ray or CT scan to check your lung function.

## Other Information

- Tell the study staff about any drugs (including prescriptions, over-the-counter drugs, or dietary supplements) you are taking or might take while you are on study.
- If you choose to take part in this research study, you must not take part in any
  other research study until your participation on this study has ended. Tell the
  study staff about any studies in which you are enrolled or may wish to enroll
  in, as there are some exceptions.

#### 2. POSSIBLE RISKS

While on this study, you are at risk for side effects. These side effects will vary from person to person. The more commonly occurring side effects are listed in this form, as are rare but serious side effects. You should discuss these with the study doctor. You may also want to ask about uncommon side effects that have been observed in small numbers of patients but are not listed in this form. Many side effects go away shortly after treatment is stopped, but in some cases side effects may be serious, long-lasting or permanent, and may even result in hospitalization and/or death.

Tell the study staff about any side effects you may have, even if you do not think they are related to the study drugs/procedures.

Imipenem-cilastatin-relebactam, cefepime, meropenem, piperacillin/tazobactam, vancomycin, daptomycin, and linezolid may each cause low blood cell counts (red blood cells, platelets, and/or white blood cells):

- A low red blood cell count (anemia) may cause difficulty breathing and/or fatigue. You may need a blood transfusion.
- A low platelet count increases your risk of bleeding (such as nosebleeds, bruising, stroke, and/or digestive system bleeding). You may need a platelet transfusion.
- A low white blood cell count increases your risk of infection (such as pneumonia and/or severe blood infection). Infections may occur anywhere and become life-threatening. Symptoms of infection may include fever, pain, redness, and difficulty breathing.

# Imipenem-Cilastatin-Relebactam Side Effects

At this time, there are no known side effects that **occur in more than 20% of patients.** 

# Occasional (occurring in 3-20% of patients)

| headache | diarrhea diarrhea | abnormal liver tests (passible liver) |
|---|---|---|
| | <ul><li>vomiting</li><li>low blood cell counts</li></ul> | (possible liver damage) |
| | (red/platelets) | |

Rare but serious (occurring in fewer than 3% of patients)

| vein inflammation | skin redness or pain | • fever |
|-------------------|----------------------|---------|
| | at infusion site | |

## Frequency not known

• diarrhea associated with *c. difficile* 

# Based on similar drugs, imipenem-cilastatin-relebactam may cause:

| central nervous system side | <ul> <li>life-threatening allergic reaction</li> </ul> |
|---|---|
| effects, including confusion or | (such as difficulty breathing, low |
| seizures | blood pressure, and/or organ |
| | failure) |

# **Cefepime Side Effects**

At this time, there are no known side effects that **occur in more than 20% of patients.** 

# Occasional (occurring in 3-20% of patients)

| skin rash | diarrhea | abnormal liver test |
|---|---|---|
| <ul> <li>low blood levels of</li> </ul> | <ul> <li>abnormal blood</li> </ul> | (possible liver |
| phosphate | test (possible | damage) |
| (possible bone | anemia) | <ul> <li>allergic reaction</li> </ul> |
| damage) | | |

# Rare but serious (occurring in fewer than 3% of patients)

| <ul> <li>hallucinations (seeing or hearing things that are not there)</li> <li>inability to speak</li> <li>seizure (which may be continuous)</li> <li>brain disease</li> <li>coma</li> <li>fever</li> <li>nervous system damage</li> </ul> | <ul> <li>abnormal salts, minerals, and/or acids in the blood (possible weakness, swelling, fatigue, low blood pressure, organ failure, heart problems, changes in mental status, and/or seizure)</li> <li>diarrhea</li> </ul> | <ul> <li>increased risk of bleeding</li> <li>low blood cell counts (white, red, platelet)</li> <li>pain and/or inflammation</li> <li>life-threatening allergic reaction (such as difficulty breathing, low blood pressure, and/or organ failure)</li> <li>infection</li> </ul> |
|---|---|---|
|---|---|---|

## Meropenem Side Effects

There are no side known side effects of meropenem that occur in more than 10% of patients.

## Exact frequency unknown but occurring in 1-10% of patients

- blood vessel disorder (possible tissue death)
- shock
- headache
- seizure
- skin rash
- low blood sugar
- nausea
- diarrhea

- vomiting
- constipation
- digestive system problems
- low red blood cells
- abnormal liver tests (possible yellowing of the skin and/or eyes)
- pain

- sore throat
- infection
- severe life-threatening infection (possible low blood pressure, kidney failure, and/or heart failure)
- injection site inflammation

## Serious side effects occurring in fewer than 1% of patients

- fast or slow heartbeat
- heart attack
- heart failure
- sudden stopping of the heart
- tissue swelling
- high blood pressure
- low blood pressure (possible dizziness/fainting)
- fever
- fainting
- hallucinations (seeing or hearing things that are not there)
- delirium (loss of contact with reality)
- allergic skin reaction
- skin rash (possible fever/lymph node swelling/inflammation of internal organs/abnormal blood cell counts)

- very severe blistering skin disease (loss of large portion of skin and/or ulcers of the skin and digestive tract)
- low blood levels of potassium (possible weakness and/or muscle cramps)
- blood in the abdomen /digestive system bleeding
- intestinal blockage
- paralysis of the intestines
- blood in the urine
- low blood cell counts (white and/or platelet)
- abnormal blood test (possible anemia)
- anemia due to destruction of red blood cells
- increased amount of blood

- low oxygen level in the blood
- abnormal bone test
- abnormal liver tests (possible liver damage)
- liver failure
- blockage of the bile tract (possible body yellowing and/or abdominal pain)
- abnormal sensation (such as pins and needles)
- chest pain
- kidney failure
- difficulty breathing (possibly due to narrowing of the airways)
- blockage in the lung (possible pain and/or shortness of breath)
- build-up of fluid around the lungs
- fluid in the lung (possible difficulty breathing)

infection

## Piperacillin/Tazobactam Side Effects

At this time, there are no known side effects that occur in more than 20% of patients.

## Occasional (occurring in 3-20% of patients)

| difficulty sleeping | • itching | upset stomach |
|---|---|---|
| <ul> <li>headache</li> </ul> | • nausea | diarrhea |
| skin rash | <ul> <li>vomiting</li> </ul> | <ul> <li>constipation</li> </ul> |

## Rare but serious (occurring in fewer than 3% of patients)

low blood pressure very severe blistering kidney inflammation (possible skin disease (loss of (possible kidney large portion of skin damage/failure) dizziness/fainting) and/or ulcers of the blood clots in a vein lung inflammation skin and digestive (possible pain, (possible difficulty swelling, and/or tract) breathing) redness) low blood sugar allergic reaction shock anemia due to life-threatening allergic destruction of red reaction (such as fever blood cells difficulty breathing, low seizures blood pressure, and/or liver damage allergic skin reaction organ failure) jaundice (yellowing of shedding and scaling skin and/or eyes) injection site reaction of the skin (possible

# Frequency Unknown

fluids)

fatal loss of bodily

low blood levels of high blood sugar high blood platelet (possible diabetes) count (possible albumin (possible swelling, weakness, increased clotting) low blood counts (red. and/or fatigue) platelet, white) abnormal liver test changes in body salts abnormal blood test (possible liver such as sodium, (possible anemia) damage) potassium, and/or increase in infectionkidney failure magnesium (possible fighting cells fatigue and/or weakness)

# **Vancomycin Side Effects**

Exact frequency unknown but occurring in more than 10% of patients

| • | low blood pressure (possible | • | skin rash on face and upper body |
|---|------------------------------|---|----------------------------------|
| | flushing/dizziness/fainting) | | |

## Exact frequency unknown but occurring in between 1 and 10% of patients

| • chills | skin rash | increase in infection- |
|----------|---------------------------------------|------------------------|
| fever | <ul> <li>vein inflammation</li> </ul> | fighting cells |
| | | low white blood cell |
| | | count |

# Exact frequency unknown but occurring in less than 1% of patients

| • | skin rash (possible | • |
|---|--------------------------|---|
| | fever/lymph node | |
| | swelling/inflammation of | |
| | internal | |
| | organs/abnormal blood | • |
| | cell counts) | |

- very severe blistering skin disease (with ulcers of the skin and digestive tract)
- low platelet cell count
- hearing loss
- kidney failure
- blood vessel inflammation (possible bleeding and/or bruising)

# **Daptomycin Side Effects**

There are currently no known side effects occurring in more than 20% of patients.

# Occasional (occurring in 3-20% of patients)

- chest pain
- swelling (arm/leg)
- high blood pressure
- low blood pressure (possible dizziness/fainting)
- difficulty sleeping
- headache
- weakness
- dizziness
- anxiety
- fever
- sweating
- skin rash
- itchina
- skin redness

- abnormal salts, minerals, and/or acids in the blood (possible weakness, swelling, fatigue, low blood pressure, organ failure, heart problems, changes in mental status, and/or seizure)
- vomiting/nausea
- abdominal pain
- upset stomach
- diarrhea
- constipation
- bacteria in the blood
- low red blood cell count

- pain
- muscle damage and/or breakdown
- kidney failure
- cough
- difficulty breathing
- build-up of fluid around the lungs
- injection site swelling, pain, and/or heat
- severe life-threatening infection (possible low blood pressure, kidney failure, and/or heart failure)

The drug may cause an increased risk of infection, such as pneumonia. This infection may occur anywhere (such as the urinary tract, bone, and vagina). It may become life-threatening. Symptoms of infection may include fever, pain, redness, and difficulty breathing.

## Rare but serious (occurring in fewer than 3% of patients)

- irregular heartbeat
- sudden stopping of the heart
- tissue swelling
- coma after anesthesia for surgery
- changes in mental status (such as hallucinations)
- very severe blistering skin disease (with ulcers of the skin and digestive system)
- severe blisters
- skin rash (possible fever/lymph node swelling/inflammation of internal organs/abnormal blood cell counts)

- jaundice (yellowing and/or darkening of the skin)
- digestive system bleeding
- increased risk of bleeding
- low blood cell count (white, platelet)
- high platelet count (possible increased clotting)
- uncontrolled movements
- breakdown of muscle tissue (possible kidney failure)
- abnormal sensation (such as pins and needles)

- nerve damage (possible numbness, pain, and/or loss of motor function)
- eye irritation
- blurry vision
- decreased kidney function
- type of pneumonia due to build-up of white blood cells (possible lung failure or death)
- allergic reaction, possible life-threatening (such as difficulty breathing, low blood pressure, and/or organ failure)

# **Linezolid Side Effects**

# Exact frequency unknown but occurring in more than 10% of patients

| <ul> <li>headache</li> </ul> | <ul><li>diarrhea</li></ul> | <ul> <li>low blood cell counts</li> </ul> |
|---|---|---|
| | | (red/white/platelets) |

# Exact frequency unknown but occurring in between 1 and 10% of patients

- feverdifficulty sleeping
- dizziness
- skin rash
- itching
- abnormal blood test (possible pancreas damage)
- abnormal blood test
- nausea
- vomiting
- abnormal digestive blood test (possible inflammation of the pancreas)
- constipation
- abnormal taste
- abdominal pain

- tongue discoloration
- inflammation of the pancreas (possible abdominal pain)
- abnormal liver tests
   (possible liver damage
   and/or possible
   yellowing of the
   skin/eyes)
- tissue swelling
- blurred vision

# Exact frequency unknown but occurring in less than 1% of patients

- high blood pressure
- nerve damage (possible numbness, pain, and/or loss of motor function)
- seizures
- large skin blisters
- very severe blistering skin disease (with ulcers of the skin and digestive tract)
- low blood sugar

- abnormal blood acid/base balance (possible organ damage)
- breakdown of muscle tissue (possible kidney failure)
- high levels of serotonin (possible seizures, muscle breakdown, headache, fast heart rate, and/or shivering/sweating)
- nerve damage (affecting the eye)
- blindness
- life-threatening allergic reaction (such as difficulty breathing, low blood pressure, and/or organ failure)

**Using the study drugs together** may cause side effects that are not seen when each is given alone. The study drug combination may also increase the frequency and/or severity of the side effects listed above.

### Other Risks

**Blood draws** may cause pain, bleeding, and/or bruising. You may faint and/or develop an infection with redness and irritation of the vein at the site where blood is drawn. Frequent blood collection may cause anemia (low red blood cell count), which may create a need for blood transfusions.

**CT scans** send x-rays through the body at many different angles. You will be exposed to a small dose of radiation. All radiation adds up over a lifetime and may increase the risk of new cancer forming. Some people may feel "closed in" while lying in the scanner. However, the scanner is open at both ends, and an intercom allows you to talk with doctors and staff. If you feel ill or anxious during scanning, doctors and/or radiology technicians will give comfort, or the scanning will be stopped. Solution may also be given by vein to make the x-ray pictures more accurate. This may cause an uncomfortable feeling of warmth, nausea, and/or severe allergic reactions. The solution injection may also cause pain, bleeding, bruising, hives, and/or itching.

**X-rays** send a small amount of radiation though the body. All radiation adds up over a lifetime and may increase the risk of a new cancer forming.

Although every effort will be made to keep study data safe, there is a chance that your personal health information could be lost or stolen, which may result in a **loss of confidentiality**.

This study may involve unpredictable risks to the participants.

#### **Pregnancy Related Risks**

Taking part in this study can result in risks to an unborn or breastfeeding baby, so you should not become pregnant, breastfeed a baby, or father a child while on this study. You must use birth control during the study and for at least 28 days after your last dose of study drugs, if you are sexually active.

Birth Control Specifications: If you can become pregnant or father a child, you must use 2 forms of birth control. Acceptable forms of birth control include either 2 barrier methods (like a condom or diaphragm with spermicide) or 1 barrier method plus a hormonal method (such as birth control pills/injections/patches).

If you have had surgery to make you sterile or you went through menopause at least 2 years ago, you do not need to use birth control while on study.

Males: Tell the doctor right away if your partner becomes pregnant or suspects pregnancy while on study or within 28 days after your last dose of study drugs. If your partner/spouse becomes pregnant while you are on this study, the sponsor would like to collect information about the pregnancy. The study sponsor's contact information will be made available so that, if you and your partner wish to, you can share information about the outcome of the pregnancy with the sponsor. If you and/or your partner choose not to share this information, it will not result in any penalty or loss of benefits to which you are otherwise entitled.

Females: If you become pregnant or suspect that you are pregnant, you must tell your doctor right away. The sponsor will ask for information about the pregnancy.

Getting pregnant will result in your removal from this study.

#### 3. COSTS AND COMPENSATION

If you suffer injury as a direct result of taking part in this study, MD Anderson health providers will provide medical care. However, this medical care will be billed to your insurance provider or you in the ordinary manner. You will not be reimbursed for expenses or compensated financially by MD Anderson or Merck for this injury. You may also contact the Chair of MD Anderson's IRB at 713-792-6477 with questions about study-related injuries. By signing this consent form, you are not giving up any of your legal rights.

Certain tests, procedures, and/or drugs that you may receive as part of this study may be without cost to you because they are for research purposes only. However, your insurance provider and/or you may be financially responsible for the cost of care and treatment of any complications resulting from the research tests, procedures, and/or drugs. Standard medical care that you receive under this research study will be billed to your insurance provider and/or you in the ordinary manner. Before taking part in this study, you may ask about which parts of the research-related care may be provided without charge, which costs your insurance

provider may pay for, and which costs may be your responsibility. You may ask that a financial counselor be made available to you to talk about the costs of this study.

Samples that are collected from you in this study may be used for the development of treatments, devices, new drugs, or patentable procedures that may result in commercial profit.

There are no plans to compensate you for any patents or discoveries that may result from your participation in this research.

You will receive no compensation for taking part in this study.

## **Additional Information**

- 4. You may ask the study chair (Dr. Issam Raad, at 713-792-6237) any questions you have about this study. You may also contact the Chair of MD Anderson's Institutional Review Board (IRB a committee that reviews research studies) at 713-792-6477 with any questions that have to do with this study or your rights as a study participant.
- 5. You may choose not to take part in this study without any penalty or loss of benefits to which you are otherwise entitled. You may also withdraw from participation in this study at any time without any penalty or loss of benefits. If you decide you want to stop taking part in the study, it is recommended for your safety that you first talk to your doctor. If you withdraw from this study, you can still choose to be treated at MD Anderson.

The study staff may ask if they can continue collecting the results of routine care from your medical record.

- 6. This study or your participation in it may be changed or stopped without your consent at any time by the study chair, Merck, the U.S. Food and Drug Administration (FDA), the Office for Human Research Protections (OHRP), or the IRB of MD Anderson.
- 7. You will be informed of any new findings or information that might affect your willingness to continue taking part in the study, including the results of all of your standard tests performed as part of this research, and you may be asked to sign another informed consent and authorization form stating your continued willingness to participate in this study.

Most tests done on samples in research studies are only for research and have no clear meaning for health care. If the research with your identifiable information or samples gives results that do have meaning for your health, the researchers will not contact you to let you know what they have found.

8. MD Anderson may benefit from your participation and/or what is learned in this

study.

- 9. This study is sponsored and/or supported by: Merck.
- 10. In a medical emergency, you may be cared for by someone who has a financial interest with the study sponsor(s)/supporter. If you have any questions about this, you may call the IRB at 713-792-6477.

#### **Future Research**

#### Data

Your personal information is being collected as part of this study. These data may be used by researchers at MD Anderson or Merck and/or shared with other researchers and/or institutions for use in future research.

#### Samples

Samples (such as blood and/or tissue) are being collected from you as part of this study. Researchers at MD Anderson may use any leftover samples that are stored at MD Anderson in future research. Leftover samples stored at Merck will not be used in future research.

If you do not want your samples or data to be used for future research, tell the study doctor. You may withdraw your samples at any time by telling your study team. If you decide to withdraw your samples, they will be returned to the lab they came from or destroyed. However, the data and test results already collected from your samples will be kept and may be used.

Before being used or shared for future research, every effort will be made to remove your identifying information from any data and/or research samples. If all identifying information is removed, you will not be asked for additional permission before future research is performed.

In some cases, all of your identifying information may not be removed before your data or research samples are used for future research. If future research is performed at MD Anderson, the researchers must get approval from the Institutional Review Board (IRB) of MD Anderson before your data and/or research samples can be used. At that time, the IRB will decide whether or not further permission from you is required. The IRB is a committee of doctors, researchers, and community members that is responsible for protecting study participants and making sure all research is safe and ethical.

If you do not want your samples or data to be used for future research, tell the study doctor. You may withdraw your samples at any time by telling your study team. If you decide to withdraw your samples, they will be returned to the lab they came from or destroyed. However, the data and test results already collected from your samples will be kept and may be used.

If this research is not performed at MD Anderson, MD Anderson will not have oversight of any data and/or samples.

#### **Genetic Research**

Research samples collected from you as part of this study will not be used for genetic research.

#### **Conflict of Interest**

Dr. Issam Raad (Study Chair) has received compensation from Merck as a Consultant. The financial interests are within the limits of the conflict of interest policy.

Dr. Ray Hachem (Study Co-Chair) has received compensation from Merck as a Speaker. The financial interests are within the limits of the conflict of interest policy.

## **Authorization for Use and Disclosure of Protected Health Information (PHI):**

- A. During the course of this study, MD Anderson will be collecting and using your PHI, including identifying information, information from your medical record, and study results. For legal, ethical, research, and safety-related reasons, your doctor and the research team may share your PHI with:
  - Federal agencies that require reporting of clinical study data (such as the FDA, National Cancer Institute [NCI], and OHRP)
  - The IRB and officials of MD Anderson
  - Merck, Inc., who is a sponsor or supporter of this study, and/or any future sponsors/supporters of the study
  - Study monitors and auditors who verify the accuracy of the information
  - Individuals who put all the study information together in report form

Study sponsors and/or supporters receive limited amounts of PHI. They may also view additional PHI in study records during the monitoring process. MD Anderson's contracts require sponsors/supporters to protect this information and limit how they may use it.

The results of this research may be published in scientific journals or presented at medical meetings, but your identity will not be disclosed.

- B. Signing this consent and authorization form is optional but you cannot take part in this study or receive study-related treatment if you do not agree and sign.
- C. MD Anderson will keep your PHI confidential when possible (according to state and federal law). However, in some situations, the FDA could be required to reveal the names of participants.

Once disclosed outside of MD Anderson, federal privacy laws may no longer protect your PHI.

- D. The permission to use your PHI will continue indefinitely unless you withdraw your authorization in writing. Instructions on how to do this can be found in the MD Anderson Notice of Privacy Practices (NPP) or you may contact the Chief Privacy Officer at 713-745-6636. If you withdraw your authorization, you will be removed from the study and the data collected about you up to that point can be used and included in data analysis. However, no further information about you will be collected.
- E. A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

# **CONSENT/AUTHORIZATION**

I understand the information in this consent form. I have had a chance to read the consent form for this study, or have had it read to me. I have had a chance to think

| permission to enroll me on this study. By signing this consent form, I any of my legal rights. I will be given a signed copy of this consent d | l am not giving up |
|---|---|
| SIGNATURE OF PARTICIPANT | DATE |
| PRINTED NAME OF PARTICIPANT | |
| WITNESS TO CONSENT I was present during the explanation of the research to be performed | under this protocol |
| SIGNATURE OF WITNESS TO THE VERBAL CONSENT PRESENTATION (OTHER THAN PHYSICIAN OR STUDY CHAIR) A witness signature is only required for non-English speakers utilizing the short form consent process (VTPS) and patients who are illiterate. | DATE |
| PRINTED NAME OF WITNESS TO THE VERBAL CONSENT | |
| PERSON OBTAINING CONSENT I have discussed this research study with the participant and/or his o representative, using language that is understandable and appropriate have fully informed this participant of the nature of this study and its pand risks and that the participant understood this explanation. | te. I believe that I |
| PERSON OBTAINING CONSENT | DATE |
| PRINTED NAME OF PERSON OBTAINING CONSENT | |
| <u>TRANSLATOR</u> | |
| I have translated the above informed consent as written (without add subtractions) intoand assisted (Name of Language) | |
| obtaining and providing consent by translating all questions and resp consent process for this participant. | oonses during the |
| NAME OF TRANSLATOR SIGNATURE OF TRANSLATOR | DATE |
| ☐ Please check here if the translator was a member of the research a witness, other than the translator, must sign the witness line.) | team. (If checked |